CLINICAL TRIAL: NCT01658488
Title: Pilot Study of the Effect of Iron Fortified Rice on Iron Stores and Reticulocytes in Iron Deficient Anemic Women
Brief Title: Pilot Study of the Effect of Iron Fortified Rice in Iron Deficient Anemic Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: The Wright Group in Crowley, LA (Unknown)
Responsible Party: Principal Investigator, Frank Greenway, Principal Investigator, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PBRC 12026
Record Dates: First submitted 2012-07-30; First posted 2012-08-07 (Estimated); Last update posted 2018-11-01 (Actual); Status verified 2018-10

CONDITIONS: Iron Deficiency Anemia
Keywords: Iron deficiency anemia; rice
MeSH Terms: conditions — Anemia, Iron-Deficiency

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Regular Rice (Other): 2 servings per day of non-fortified rice
  Interventions: Other: Non-fortified rice
- Iron-fortified Rice (Other): 2 servings per day of Rice enriched in iron for women with iron-deficient anemia to restore their blood counts more efficiently than the standard rice not enriched with iron.
  Interventions: Other: Iron-fortified Rice

INTERVENTIONS:
Other: Non-fortified rice — Consumption of 2 servings of Non-fortified rice per day in women with iron deficiency anemia and measure serum iron and transferrin at baseline and end of study.
  Arms: Regular Rice
Other: Iron-fortified Rice — Consumption of 2 servings of Iron-fortified rice per day in women with iron deficiency anemia and measure serum iron and transferrin at baseline and end of study.
  Arms: Iron-fortified Rice

SUMMARY:
The purpose of this study is to see if rice enriched in iron will help women with iron-deficient anemia restore their blood counts more efficiently than the standard rice not enriched with iron.

DETAILED DESCRIPTION:
The study will consist of 1 screening visit and 3 study visits. The two-week study will be scheduled to be between menses.

You will then be assigned to eat regular rice dishes or rice dishes fortified with iron for the two-week period. The assignment to the rice group will be made randomly (like flipping a coin). Your chance of being in either rice group will be 50:50. You will be given 14 frozen rice meals in styrofoam containers to take home. You will be expected to eat two rice dishes per day for the next study week and to bring the empty containers to your next study visit.

ELIGIBILITY:
Inclusion Criteria:

* Are a healthy woman.
* Are between 18 and 50 years of age.
* Have iron deficient anemia.

Exclusion Criteria:

* Are pregnant or nursing.
* Are taking a medication or supplement to treat iron deficiency.
* Treatment for iron deficiency within the past month
* Type 1 or type 2 diabetes
* Ongoing cancer
* Active auto-immune disease
* Chronic infections (e.g. HIV/AIDS, hepatitis B, hepatitis C)
* Chronic kidney disease
* Liver cirrhosis
* History of drug or alcohol abuse within the past 6 months
* History of eating disorder within the past 6 months
* Any gastrointestinal surgery affecting nutrient absorption

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2012-07; Primary Completion 2015-08 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change in reticulocyte count. | Baseline and 1 and 2 weeks following consumption of 2 servings
  Change in reticulocyte typically count in the iron-fortified rice group compared to the regular rice group. This is a test that measures how rapidly immature red blood cells called reticulocytes are made by the bone marrow and released into the blood.

SECONDARY OUTCOMES:
Changes in serum iron | Baseline and 1 and 2 weeks following consumption
  Changes in serum iron is a medical laboratory test that measures the amount of circulating iron in the blood; in the fortified rice group compared to the regular rice group.
Transferrin | Baseline and 1 and 2 weeks following consumption
  Changes in transferrin (a protein that transports iron in the body ) in the fortified rice group compared to the regular rice group.
Hemoglobin | Baseline and 1 and 2 weeks following consumption
  Changes in hemoglobin (The key protein in red blood cells to which oxygen attaches) in the fortified rice group compared to the regular rice group.
Hematocrit | Baseline and 1 and 2 weeks following consumption
  Changes in hematocrit (the proportion of your total blood volume that is composed of red blood cells) in the fortified rice group compared to the regular rice group.
Mean Corpuscular Volume | Baseline and 1 and 2 weeks following consumption
  Changes in mean corpuscular volume (the average red blood cell size in the fortified rice group compared to the regular rice group.

CONTACTS AND LOCATIONS:
Overall Officials: Frank L. Greenway, MD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

REFERENCES:
- [Result] Losso JN, Karki N, Muyonga J, Wu Y, Fusilier K, Jacob G, Yu Y, Rood JC, Finley JW, Greenway FL. Iron retention in iron-fortified rice and use of iron-fortified rice to treat women with iron deficiency: A pilot study. BBA Clin. 2017 Sep 8;8:78-83. doi: 10.1016/j.bbacli.2017.09.001. eCollection 2017 Dec. PMID 28966915